CLINICAL TRIAL: NCT03798054
Title: A Randomized, 24 Week, Active-controlled, Open-label, 3-arm, Parallel-group Multicenter Study Comparing the Efficacy and Safety of iGlarLixi to Insulin Glargine and Lixisenatide in Type 2 Diabetes Mellitus Patients Insufficiently Controlled With Oral Antidiabetic Drug(s)
Brief Title: Evaluation of Insulin Glargine/Lixisenatide Fixed Ratio Combination in Patients With Type 2 Diabetes Insufficiently Controlled With Oral Antidiabetic Drug(s)
Acronym: Lixilan-O-AP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14943; U1111-1190-7669 (Other: UTN)
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Metformin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Soliqua (insulin glargine/lixisenatide) (Experimental): iGlarLixi (insulin glargine/lixisenatide) will be self-administered subcutaneously once daily in the morning on top of metformin for 24 weeks.
  Interventions: Drug: Insulin glargine/Lixisenatide (HOE901/AVE0010); Drug: Metformin; Drug: SGLT2 inhibitor
- Lantus (insulin glargine) (Active Comparator): Insulin glargine will be self-administered subcutaneously once daily at any time of the day on top of metformin for 24 weeks. Injection time should be determined on the day of randomization, and should remain about the same until the end of the treatment period.
  Interventions: Drug: Insulin glargine (HOE901); Drug: Metformin; Drug: SGLT2 inhibitor
- Lyxumia (lixisenatide) (Active Comparator): Lixisenatide will be self-administered subcutaneously once daily according to the locally approved label on top of metformin for 24 weeks. Injection time should be determined on the day of randomization, and should remain about the same until the end of the treatment period.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Metformin; Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: Insulin glargine/Lixisenatide (HOE901/AVE0010) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Soliqua; iGlarLixi
  Arms: Soliqua (insulin glargine/lixisenatide)
Drug: Insulin glargine (HOE901) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Lantus
  Arms: Lantus (insulin glargine)
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Lyxumia
  Arms: Lyxumia (lixisenatide)
Drug: Metformin — Pharmaceutical form: tablet
  Route of administration: oral
Drug: SGLT2 inhibitor — Pharmaceutical form:tablet
  Route of administration: oral

SUMMARY:
Primary Objectives:

The co-primary objective of this study is:

* To demonstrate the superiority of iGlarLixi (fixed ratio combination of insulin glargine and lixisenatide) versus lixisenatide on glycemic control as assessed by glycated hemoglobin A1c (HbA1c) change.
* To demonstrate the non-inferiority of iGlarLixi versus insulin glargine on glycemic control as assessed by HbA1c change.

Secondary Objectives:

* To assess the effects of iGlarLixi in comparison with insulin glargine alone and lixisenatide alone.
* To assess the safety in each treatment group.

DETAILED DESCRIPTION:
The maximum study duration per patient will be approximately 31 weeks: an up-to 6-week screening and run-in period (with an up-to 2-week screening phase and a 4-week run-in phase), followed by a 24-week randomized treatment period and a 3-day post-treatment safety follow up period.

ELIGIBILITY:
Inclusion criteria :

* Patients with type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year before the screening visit (V1), treated for at least 3 months prior to the screening visit (V1) with metformin alone or metformin and a second oral antidiabetic treatment that can be a sulfonylurea (SU), a glinide, an alpha-glucosidase inhibitor (alpha-GI), a dipeptidyl peptidase-4 (DPP-4) inhibitor or a sodium-glucose co transporter 2 (SGLT-2) inhibitor and who are not adequately controlled with this treatment.
* Signed written informed consent.

Exclusion criteria:

* Age < legal age of majority at the screening visit (V1).
* Body mass index (BMI) >40 kg/m² at screening.
* Glycated hemoglobin A1c (HbA1c) at screening visit:
* <7.5% or >11% for patients previously treated with metformin alone;
* <7.0% or >10% for patients previously treated with metformin and a second oral antidiabetic treatment.
* History of hypoglycemia unawareness.
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening.
* Use of oral or injectable glucose-lowering agents other than those stated in the inclusion criteria within 3 months prior to screening.
* Previous treatment with insulin (except for short-term treatment due to intercurrent illness at the discretion of the Investigator) within 1 year prior to screening.
* History of discontinuation of a previous treatment with glucagon-like-peptide-1 receptor agonists (GLP-1 RAs) due to safety/tolerability reasons or lack of efficacy.
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to screening.
* Use of weight loss drugs within 3 months prior to screening.
* Use of any investigational drug other than specified in this protocol within 1 month or 5 half-lives, whichever is longer, prior to screening.
* Within 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization.
* Planned coronary, carotid, or peripheral artery revascularization procedures to be performed during the study period.
* Known history of drug or alcohol abuse within 6 months prior to screening.
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic blood pressure >180 mmHg or diastolic blood pressure >95 mmHg.
* Laboratory findings at screening visit (V1):
* Amylase and/or lipase >3 times the upper limit of normal (ULN) laboratory range.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 ULN.
* Total bilirubin >1.5 ULN (except in case of Gilbert's syndrome).
* Calcitonin ≥20 pg/mL (5.9 pmol/L).
* Hemoglobin <10.5 g/dL and/or neutrophils <1500/mm3 and/or platelets <100 000/mm3.
* Positive urine pregnancy test in female of childbearing potential.
* Patient who has a severe renal function impairment with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 or end-stage renal disease.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy has been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (eg, multiple endocrine neoplasia syndromes).
* Use of SU, glinide, alpha-GI, DPP-4 inhibitor, and SGLT-2 inhibitor after start of run-in (from V2 [Week -4]).
* HbA1c at V4 (Week -1) : <7.0% or >10%.
* Fasting plasma glucose >250 mg/dL (13.9 mmol/L) at V4 (Week-1) (can be repeated once to confirm).
* Metformin maximal tolerated dose <1500 mg/day.
* Amylase and/or lipase >3 ULN at V4 (Week-1).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From Baseline to Week 24
  Change in glycated hemoglobin (HbA1c) from baseline to Week 24

SECONDARY OUTCOMES:
Change in postprandial plasma glucose (PPG) | From Baseline to Week 24
  Absolute change in 2-hour blood glucose excursion and PPG during meal test from baseline to Week 24 (for all patients in iGlarLixi or insulin glargine group and patients who receive morning injection in the lixisenatide group)
Change in fasting plasma glucose (FPG) | From Baseline to Week 24
  Absolute change in FPG from baseline to Week 24
Change in self-monitored plasma glucose (SMPG) profile | From Baseline to Week 24
  Absolute change in 7-point SMPG profiles from baseline to Week 24 (each time point and average daily value)
Patients with HbA1c <7.0% | At Week 24
  Percentage of patients reaching HbA1c <7% at Week 24
Patients with HbA1c ≤ 6.5% | At Week 24
  Percentage of patients reaching HbA1c ≤ 6.5% at Week 24
Change in body weight | From Baseline to Week 24
  Absolute change in body weight from baseline to Week 24
Patients with HbA1c <7.0% with no body weight gain | At Week 24
  Percentage of patients reaching HbA1c <7% with no body weight gain at Week 24
Patients with HbA1c <7.0% with no body weight gain and no documented symptomatic hypoglycemia | At Week 24
  Percentage of patients reaching HbA1c <7% with no body weight gain at Week 24 and no documented (plasma glucose [PG] ≤70 mg/dL [3.9 mmol/L]) symptomatic hypoglycemia during the 24 week treatment period
Confirmed hypoglycemia | From Baseline to Week 24
  Including severe hypoglycemia and episodes of hypoglycemia documented with PG ≤70 mg/dL (3.9 mmol/L) regardless of symptoms from baseline to Week 24
Adverse events (AEs) | From Baseline to Week 24
  Number of AEs, serious AEs, AEs of Special Interest, and AEs requiring specific monitoring from baseline to Week 24
Immunogenicity (antibody variables) | From Baseline to Week 24
  Anti-lixisenatide antibodies and anti-insulin antibodies (depending on the treatment group) from baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (79):
- China (59):
  - Investigational Site Number 1560001, Beijing
  - Investigational Site Number 1560006, Beijing
  - Investigational Site Number 1560049, Beijing
  - Investigational Site Number 1560039, Cangzhou
  - Investigational Site Number 1560009, Changchun
  - Investigational Site Number 1560027, Changchun
  - Investigational Site Number 1560016, Changsha
  - Investigational Site Number 1560053, Chengdu
  - Investigational Site Number 1560056, Chengdu
  - Investigational Site Number 1560010, Chenzhou
  - Investigational Site Number 1560037, Chongqing
  - Investigational Site Number 1560050, Chongqing
  - Investigational Site Number 1560044, Dongguan
  - Investigational Site Number 1560033, Guangzhou
  - Investigational Site Number 1560028, Guangzhou
  - Investigational Site Number 1560012, Handan
  - Investigational Site Number 1560023, Hangzhou
  - Investigational Site Number 1560035, Harbin
  - Investigational Site Number 1560036, Harbin
  - Investigational Site Number 1560011, Hengshui
  - Investigational Site Number 1560024, Hohhot
  - Investigational Site Number 1560047, Hohhot
  - Investigational Site Number 3440001, Hong Kong
  - Investigational Site Number 1560026, Huanggang
  - Investigational Site Number 1560025, Huangshi
  - Investigational Site Number 1560048, Huizhou
  - Investigational Site Number 1560034, Huzhou
  - Investigational Site Number 1560005, Jinan
  - Investigational Site Number 1560052, Jinhua
  - Investigational Site Number 1560031, Jinzhou
  - Investigational Site Number 1560022, Nanjing
  - Investigational Site Number 1560014, Nanjing
  - Investigational Site Number 1560043, Nanjing
  - Investigational Site Number 1560041, Nanning
  - Investigational Site Number 1560032, Qingdao
  - Investigational Site Number 1560038, Qinhuangdao
  - Investigational Site Number 1560013, Shanghai
  - Investigational Site Number 1560007, Shanghai
  - Investigational Site Number 1560004, Shanghai
  - Investigational Site Number 1560029, Shanghai
  - Investigational Site Number 1560003, Shenyang
  - Investigational Site Number 1560054, Shenzhen
  - Investigational Site Number 1560019, Suzhou
  - Investigational Site Number 1560059, Suzhou
  - Investigational Site Number 1560021, Tianjin
  - Investigational Site Number 1560017, Tianjin
  - Investigational Site Number 1560058, Ürümqi
  - Investigational Site Number 1560018, Wuhan
  - Investigational Site Number 1560008, Xi'an
  - Investigational Site Number 1560055, Xi'an
  - Investigational Site Number 1560051, Xingtai
  - Investigational Site Number 1560030, Xining
  - Investigational Site Number 1560040, Yanji
  - Investigational Site Number 1560060, Yueyang
  - Investigational Site Number 1560046, Yueyang
  - Investigational Site Number 1560045, Zhengzhou
  - Investigational Site Number 1560002, Zhenjiang
  - Investigational Site Number 1560015, Zhuzhou
  - Investigational Site Number 1560057, Zigong
- Malaysia (6):
  - Investigational Site Number 4580001, Kelantan
  - Investigational Site Number 4580005, Kuala Lumpur
  - Investigational Site Number 4580003, Kuala Lumpur
  - Investigational Site Number 4580006, Kuching
  - Investigational Site Number 4580002, Putrajaya
  - Investigational Site Number 4580004, Seremban
- South Korea (11):
  - Investigational Site Number 4100009, Ansan-si
  - Investigational Site Number 4100012, Busan
  - Investigational Site Number 4100010, Guri-Si, Gyeonggi-Do
  - Investigational Site Number 4100004, Gwangju
  - Investigational Site Number 4100003, Seongnam-si
  - Investigational Site Number 4100016, Seoul
  - Investigational Site Number 4100011, Seoul
  - Investigational Site Number 4100013, Seoul
  - Investigational Site Number 4100001, Seoul
  - Investigational Site Number 4100002, Seoul
  - Investigational Site Number 4100005, Wŏnju
- Taiwan (3):
  - Investigational Site Number 1580003, Taichung
  - Investigational Site Number 1580005, Tainan Hsien
  - Investigational Site Number 1580004, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Yang W, Dong X, Li Q, Cheng Z, Yuan G, Liu M, Xiao J, Gu S, Niemoeller E, Chen L, Ping L, Souhami E; LixiLan-O-AP trial investigators. Efficacy and safety benefits of iGlarLixi versus insulin glargine 100 U/mL or lixisenatide in Asian Pacific people with suboptimally controlled type 2 diabetes on oral agents: The LixiLan-O-AP randomized controlled trial. Diabetes Obes Metab. 2022 Aug;24(8):1522-1533. doi: 10.1111/dom.14722. Epub 2022 May 12. PMID 35441412
- [Derived] Guo X, Yang W, Zhang J, Dong X, Liu M, Gu S, Lauand F, Li L, Huang Q, Kang L, Souhami E. iGlarLixi provides a higher derived time-in-range versus insulin glargine 100 U/mL or lixisenatide in Asian Pacific people with type 2 diabetes: A post hoc analysis. Diabetes Obes Metab. 2023 Jul;25(7):2005-2011. doi: 10.1111/dom.15074. Epub 2023 May 3. PMID 36999231